CLINICAL TRIAL: NCT07231302
Title: Determination of Stereotactic Landmarks Based on Computer-generated Images and Electrophysiological Recording Patterns for Electrode Implantation for Stimulation of the Dentate Nucleus and Its Fiber Projections Aiming the Treatment of Movement Disorders, Like Secondary Dystonia, Ataxia, Tremor (Essential and Symptomatic)
Brief Title: Stimulation of the Dentate Nucleus of the Cerebellum for the Treatment of Refractory Spasticity With or Without Dystonia
Acronym: DN_DBS
Status: Completed | Type: Observational
Sponsor: Kleber Paiva Duarte (Other)
Responsible Party: Sponsor-Investigator, Kleber Paiva Duarte, assistant professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: 32779514.5.0000.0068
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Ataxia - Other; Dystonia Disorder; Tremor, Essential; Choreatic Disorder; Deep Brain Stimulation Surgery
Keywords: Deep brain stimulation; Nucleus dentatus; Dystonia; Ataxia
MeSH Terms: conditions — Dystonic Disorders; Essential Tremor; Chorea; Dystonia; Ataxia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Final Stereotactics coordinates in DN-DBS: Computational dataset
  Interventions: Other: Analytical observation

INTERVENTIONS:
Other: Analytical observation — Analysts observation; CT + MRI + DTI pre and post operative stereotactic coordinates - implants DBS in DN

SUMMARY:
Electrical stimulation (DBS) through electrodes implanted in the dentate nucleus of the cerebellum for the treatment of tremor intractable with medication, dystonia due to cerebrovascular disease (stroke), sequelae of traumatic brain injury, and ataxia (a disease that causes incoordination of movements). Use of advanced magnetic resonance imaging techniques and recording of nerve cell activity in this nucleus

DETAILED DESCRIPTION:
To establish anatomical and functional criteria, based on stereotactic imaging and electrophysiological recordings, that enable the precise implantation of electrodes in the DN and its efferent projections for the treatment of movement disorders. This study aims to describe a surgical technique for the implantation of deep brain electrodes targeting the stimulation (DBS) of the dentate nucleus (DN) and its efferent projections, supported by the magnetic resonance imaging (MRI), the diffusion tensor imaging (DTI), reformatted in the stereotomographic images and related to stereotactic landmarks and checked with semimicro deep brain recording.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Clinical diagnosis of cerebellar syndrome resulting from stroke and spinocerebellar degeneration, intractable tremor, primary or secondary dystonia, refractory to drug and physiotherapy treatment;
3. Signed the term of free and informed consent

Exclusion Criteria:

1. Age under 18 years;
2. Presence of severe anatomical deformities in the cerebellum and/or brainstem;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dystonia, ataxia or tremor
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
DSB in the dentate nucleus | From enrollment to the end of treatment at 16 weeks
  All stereotactic image calculations the definitive location of the implants in relation to the targets proposed in the ND, were reanalyzed in a digital environment that included co-registration of the preoperative MRI, DTI, and stereotomograph

IPD SHARING:
Plan to Share IPD: Undecided
There are other projects similar to this one underway. I'd like to be able to connect with other researchers and share our challenges and findings.

REFERENCES:
- [Result] Diniz JM, Cury RG, Iglesio RF, Lepski GA, Franca CC, Barbosa ER, de Andrade DC, Teixeira MJ, Duarte KP. Dentate nucleus deep brain stimulation: Technical note of a novel methodology assisted by tractography. Surg Neurol Int. 2021 Aug 9;12:400. doi: 10.25259/SNI_338_2021. eCollection 2021. PMID 34513166